CLINICAL TRIAL: NCT00753415
Title: A Phase I Investigation of the Safety, Tolerability and Immunogenicity of V934/V935 hTERT Vaccination in Cancer Patients With Selected Solid Tumors
Brief Title: A Study of V934/V935 Vaccine in Cancer Participants With Selected Solid Tumors (V934-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V934-002; 2008_541 (Other: Merck Registration Number (Telerx #))
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Non-Small Cell Lung Carcinoma; Breast Cancer; Melanoma; Upper GI Tract Carcinoma; Colon Carcinoma; Renal Cell Carcinoma; Bladder Carcinoma; Prostate Cancer
Keywords: Urinary Bladder Neoplasms; Breast Neoplasms; Renal Cell carcinoma; Melanoma; Prostatic Neoplasms; Colonic Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Urinary Bladder Diseases; Urologic Diseases; Breast Diseases; Skin Diseases; Neoplasms; Glandular and Epithelial Neoplasms by Histologic Type; Adenocarcinoma; Kidney Neoplasms; Kidney Diseases; Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms, Nerve Tissue; Nevi and Melanomas; Genital Neoplasms; Male Genital Diseases; Male, Prostatic Diseases; Colorectal Neoplasms; Intestinal Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Melanoma; Colonic Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Prostatic Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Urinary Bladder Diseases; Urologic Diseases; Breast Diseases; Skin Diseases; Neoplasms; Adenocarcinoma; Kidney Neoplasms; Kidney Diseases; Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms, Nerve Tissue; Nevi and Melanomas; Genital Diseases, Male; Prostatic Diseases; Colorectal Neoplasms; Intestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Part A: V935 LD (Experimental): Two intramuscular (IM) injections of V935 low dose (LD), 1 given every other week over a 3-week period.
  Interventions: Biological: V935
- Part A: V934 LD(3)+V935 LD (Experimental): Three electroporation (EP) injections of V934 (LD) , 1 given every other week over a 5-week period. Following a 4-week observation period, 2 IM injections of V935 (LD) will be administered, 1 given every other week over a 3-week period.
  Interventions: Biological: V935; Biological: V934-EP
- Part A: V935 HD (Experimental): Two IM injections of V935 high dose (HD), 1 given very other week over a 3-week period.
  Interventions: Biological: V935
- Part A: V934 HD(3)+V935 HD (Experimental): Three EP injections of V934 (HD), 1 given every other week over a 5-week period. Following a 4-week observation period, 2 IM injections of V935 (HD) will be administered, 1 given every other week over a 3-week period.
  Interventions: Biological: V935; Biological: V934-EP
- Part A: V934 HD(5)+V935 HD (Experimental): Five EP injections of V934 (HD), 1 given every other week over a 9-week period. Following a 4-week observation period, 2 IM injections of V935 (HD) will be administered, 1 given every other week over a 3-week period.
  Interventions: Biological: V935; Biological: V934-EP
- Part B: V935 LD/V934 Booster (Experimental): Participants who completed Part A could enter Part B. Following a 12-week observation period, 3 EP injections of V934 booster were administered, 1 given every 2 weeks.
  Interventions: Biological: V934-EP
- Part B: V934 LD(3)+V935 LD/V934 Booster (Experimental): Participants who complete Part A can enter Part B. Following a 12-week observation period, 3 EP injections of V934 booster will be administered, 1 given every 2 weeks.
  Interventions: Biological: V934-EP
- Part B: V935 HD/V934 Booster (Experimental): Participants who complete Part A can enter Part B. Following a 12-week observation period, 3 EP injections of V934 booster will be administered, 1 given every 2 weeks.
  Interventions: Biological: V934-EP
- Part B: V934 HD(3)+V935 HD/V934 Booster (Experimental): Participants who complete Part A can enter Part B. Following a 12-week observation period, 3 EP injections of V934 booster will be administered, 1 given every 2 weeks.
  Interventions: Biological: V934-EP
- Part B: V934 HD(5)+V935 HD/V934 Booster (Experimental): Participants who complete Part A can enter Part B. Following a 12-week observation period, 3 EP injections of V934 booster will be administered, 1 given every 2 weeks.
  Interventions: Biological: V934-EP

INTERVENTIONS:
Biological: V935 — A 0.5 mL vaccine administered IM every 2 weeks as either a LD (1 x 10^9 vector genomes/mL) or a HD (1 x 10^11 vector genomes/mL).
  Arms: Part A: V934 HD(3)+V935 HD; Part A: V934 HD(5)+V935 HD; Part A: V934 LD(3)+V935 LD; Part A: V935 HD; Part A: V935 LD
Biological: V934-EP — A 0.5 mL vaccine administered by EP as either a LD (0.5 mg plasmid/mL) or a HD (5.0 mg plasmid/mL).
  Arms: Part A: V934 HD(3)+V935 HD; Part A: V934 HD(5)+V935 HD; Part A: V934 LD(3)+V935 LD; Part B: V934 HD(3)+V935 HD/V934 Booster; Part B: V934 HD(5)+V935 HD/V934 Booster; Part B: V934 LD(3)+V935 LD/V934 Booster; Part B: V935 HD/V934 Booster; Part B: V935 LD/V934 Booster

SUMMARY:
This is a two-part study to test the safety, tolerability, and immune response for V934/V935 vaccine using a new prime-boost regimen in participants with selected solid tumors.

DETAILED DESCRIPTION:
Two vaccines will be administered: V934-electroporation (EP) either low dose (LD) or high dose (HD), and V935 either LD or HD. In Part A, participants will be assigned to V935 vaccine alone or in combination with V934-EP. Part B will be an optional part of the study, offering V934-EP vaccine booster to participants who were enrolled in Part A.

ELIGIBILITY:
Inclusion Criteria Part A

* Participant has one of the selected solid tumors with no distant metastases, and is more than 8 weeks from completion of definitive therapy with intention to cure. Selected Solid Tumors: Stage I to III non-small cell lung carcinoma (NSCLC); Stage III breast cancer; Stage IIB or III melanoma; Stage II or III upper gastrointestinal tract carcinoma (e.g., esophagus, stomach, gallbladder, pancreas); Stage III colon carcinoma; Stage II, III, or IV (M0 only) renal cell carcinoma; Stage II, III, or IV (M0 only) bladder carcinoma; clinically-localized prostate carcinoma
* Participant has adequate organ function.
* Female participant of childbearing potential has a negative serum pregnancy test within 3 days of study enrollment.

Exclusion Criteria Part A

* Participant has known hypersensitivity to any component of study vaccine.
* Participant has a history of clinically significant cardiac conditions, including cardiac arrhythmias which have not been controlled within the last 3 months, unstable angina, myocardial infarction (within the last 3 months), or New York Heart Association (NYHA) Class III or IV congestive heart failure. Participant must have no clinically significant electrocardiogram (ECG) abnormalities and not have a pacemaker or cardioverter/defibrillator implanted.
* Participant has undergone splenectomy or has any history of autoimmune disorder.
* Participant has received immunosuppressive treatment within 1 month prior to enrollment.
* Participant has known acquired, inherited, or idiopathic thrombocytopenia, platelet dysfunction or coagulopathy that would contraindicate IM injections.
* Participant has an acute infection requiring intravenous antibiotic, antiviral or antifungal agents within 2 weeks of study entry.
* Participant is pregnant or breastfeeding, or expecting to conceive at any time during the study or within 1 year after receiving the last vaccination.
* Participant is known to be Human Immunodeficiency Virus (HIV)-seropositive.
* Participant has known history of Hepatitis B or C or active Hepatitis A.
* Participant has been vaccinated for any disease or for prophylaxis within 1 month prior to the first vaccination.
* The participant has been diagnosed with Systemic Lupus Erythematosus (SLE)

Inclusion Criteria Part B

* Participant must have completed their respective vaccination Treatment Group regimen for Part A of this study.
* Participant must have completed a ≥12 week safety observation period prior to receiving their first V934-EP boost.

Exclusion Criteria Part B

* Participant has new or metastatic tumor lesions since enrollment in Part A.
* Participant has developed any significant cardiac conditions since enrollment in Part A including cardiac arrhythmias which have not been controlled within the last 3 months, unstable angina, myocardial infarction (within the last 3 months), or NYHA Class III or IV congestive heart failure.
* Participant has undergone a splenectomy, or has developed any autoimmune disorders, since enrollment in Part A.
* Participant has received immunosuppressive treatment within 1 month prior to enrollment in Part B
* Participant has developed any acquired, inherited, or idiopathic thrombocytopenia, platelet dysfunction or coagulopathy that would contraindicate IM injections
* Participant has an acute infection requiring intravenous antibiotic, antiviral or antifungal agents within 2 weeks of entry to Part B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

REFERENCES:
- [Derived] Aurisicchio L, Fridman A, Mauro D, Sheloditna R, Chiappori A, Bagchi A, Ciliberto G. Safety, tolerability and immunogenicity of V934/V935 hTERT vaccination in cancer patients with selected solid tumors: a phase I study. J Transl Med. 2020 Jan 30;18(1):39. doi: 10.1186/s12967-020-02228-9. PMID 32000810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: V935 alone or in combination with V934 was administered to 37 participants with selected solid tumors in Part A.
Pre-assignment Details: Of the 37 participants who were enrolled in Part A, 32 participants completed and were eligible to enroll in the optional extension study Part B. There were 28 participants who elected to enroll in Part B.
Groups:
- Part A: V934 LD(3)+V935 LD: Three electroporation (EP) injections of V934 (LD) were administered, 1 given every other week over a 5-week period. Following a 4-week observation period, 2 IM injections of V935 (LD) were administered, 1 given every other week over a 3-week period.
- Part A: V935 HD: Two IM injections of V935 high dose (HD), 1 given every other week over a 3-week period.
- Part A: V934 HD(3)+V935 HD: Three EP injections of V934 (HD) were administered, 1 given every other week over a 5-week period. Following a 4-week observation period, 2 IM injections of V935 (HD) were administered, 1 given every other week over a 3-week period.
- Part A: V934 HD(5)+V935 HD: Five EP injections of V934 (HD) were administered, 1 given every other week over a 9-week period. Following a 4-week observation period, 2 IM injections of V935 (HD) were administered, 1 given every other week over a 3-week period.
- Part B: V935 LD/V934 Booster: Participants who completed Part A could enter Part B. Following a 12-week observation period, 3 EP injections of V934-EP booster were administered, 1 given every 2 weeks.
- Part B: V934 LD(3)+V935 LD/V934 Booster; Part B: V935 HD/V934 Booster; Part B: V934 HD(3)+V935 HD/V934 Booster; Part B: V934 HD(5)+V934 HD/V934 Booster: Participants who completed Part A could enter Part B. Following a 12-week observation period, 3 EP injections of V934 booster were administered, 1 given every 2 weeks.
Period: Part A
Arm/Group | Part A: V935 LD | Part A: V934 LD(3)+V935 LD | Part A: V935 HD | Part A: V934 HD(3)+V935 HD | Part A: V934 HD(5)+V935 HD | Part B: V935 LD/V934 Booster | Part B: V934 LD(3)+V935 LD/V934 Booster | Part B: V935 HD/V934 Booster | Part B: V934 HD(3)+V935 HD/V934 Booster | Part B: V934 HD(5)+V934 HD/V934 Booster
Started | 3 | 3 | 10 | 11 | 10 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 8 | 9 | 10 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: V935 LD | Part A: V934 LD(3)+V935 LD | Part A: V935 HD | Part A: V934 HD(3)+V935 HD | Part A: V934 HD(5)+V935 HD | Part B: V935 LD/V934 Booster | Part B: V934 LD(3)+V935 LD/V934 Booster | Part B: V935 HD/V934 Booster | Part B: V934 HD(3)+V935 HD/V934 Booster | Part B: V934 HD(5)+V934 HD/V934 Booster
Started | 0 | 0 | 0 | 0 | 0 | 1 (Of 2 eligible participants who completed Part A, 1 chose to enter Part B) | 2 (Of 3 eligible participants who completed Part A, 2 chose to enter Part B) | 7 (Of 8 eligible participants who completed Part A, 7 chose to enter Part B) | 9 (9 participants who completed Part A were eligible and enrolled in Part B) | 9 (Of 10 eligible participants who completed Part A, 9 chose to enter Part B)
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A: V935 LD: Two IM injections of V935 low dose (LD), 1 given every other week over a 3-week period.
- Part A: V934 LD(3)+V935 LD: Three electroporation (EP) injections of V934 (LD) were administered, 1 given every other week over a 5-week period. Following a 4 week observation period, 2 IM injections of V935 (LD) were administered, 1 given every other week over a 3-week period.
- Part A: V934 HD(3)+V935 HD: Three EP injections of V934 (HD) were administered, 1 given every other week over a 5-week period. Following a 4 week observation period, 2 IM injections of V935 (HD) were administered, 1 given every other week over a 3-week period.
- Total: Total of all reporting groups
Arm/Group | Part A: V935 LD | Part A: V934 LD(3)+V935 LD | Part A: V935 HD | Part A: V934 HD(3)+V935 HD | Part A: V934 HD(5)+V935 HD | Total
Number analyzed (Participants) | 3 | 3 | 10 | 11 | 10 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.0 (9.5) | 70.0 (6.2) | 63.8 (10.0) | 58.8 (11.7) | 60.2 (11.7) | 62.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 4 | 1 | 10
  Male | 3 | 2 | 6 | 7 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLT was defined as a vaccine- or EP-related adverse event (AE) including the following: Hematological (Grade 3 neutropenia with fever, Grade 4 neutropenia ≥5 days, Grade 4 thrombocytopenia) or non-hematological AE, Grade 3, 4 or 5 with the exception of Grade 3 nausea, vomiting, diarrhea or serum glutamic oxaloacetic transaminase (SGOT) elevation, alopecia, Grade 3/4 creatinine phosphokinase (CPK) elevation or inadequately treated hypersensitivity. Any Grade 3/4 related AE that failed to return to ≤Grade 1 or baseline within 14 days was also considered a DLT.
Time Frame: Day 1 up to 30 days following the last vaccination (up to 77 weeks); Treatment Period + Acute Follow-up (FU) Period
Population: Evaluable patients who completed all scheduled vaccinations were included in the DLT analysis.
Measure: Number; unit: Participants
Groups:
- Part B: V934 HD(5)+V935 HD/V934 Booster: Participants who completed Part A could enter Part B. Following a 12-week observation period, 3 EP injections of V934 booster were administered, 1 given every 2 weeks.
Arm/Group | Part A: V935 LD | Part A: V934 LD(3)+V935 LD | Part A: V935 HD | Part A: V934 HD(3)+V935 HD | Part A: V934 HD(5)+V935 HD | Part B: V935 LD/V934 Booster | Part B: V934 LD(3)+V935 LD/V934 Booster | Part B: V935 HD/V934 Booster | Part B: V934 HD(3)+V935 HD/V934 Booster | Part B: V934 HD(5)+V935 HD/V934 Booster
Number analyzed (Participants) | 3 | 3 | 10 | 11 | 10 | 1 | 2 | 7 | 9 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: This analysis includes the number of participants with AEs and serious AEs (SAEs) during the Treatment Period plus the Acute Follow-up (FU) Period (up to 30 days following last vaccination). An AE was defined as any unfavorable or unintended change in the structure, function or chemistry of the body temporally associated with the use of the product, whether or not considered related to the product, including any worsening of a preexisting condition which was temporally associated with the product. An SAE was defined as an AE resulting in death, was life-threatening, resulted in or prolonged hospitalization, was a congenital anomaly, a cancer, an overdose or other important medical event.
Time Frame: Day 1 up to 30 days following the last vaccination (up to 77 weeks); Treatment Period + Acute Follow-up (FU) Period
Population: All Participants as Treated (APaT) population; all participants who received at least one vaccination.
Measure: Number; unit: Participants
Arm/Group | Part A: V935 LD | Part A: V934 LD(3)+V935 LD | Part A: V935 HD | Part A: V934 HD(3)+V935 HD | Part A: V934 HD(5)+V935 HD | Part B: V935 LD/V934 Booster | Part B: V934 LD(3)+V935 LD/V934 Booster | Part B: V935 HD/V934 Booster | Part B: V934 HD(3)+V935 HD/V934 Booster | Part B: V934 HD(5)+V935 HD/V934 Booster
Number analyzed (Participants) | 3 | 3 | 10 | 11 | 10 | 1 | 2 | 7 | 9 | 9
Participants | 3 | 3 | 8 | 11 | 10 | 1 | 1 | 3 | 8 | 7

3. Secondary Outcome: Number of Participants With Immunologic Response to V934/V935 (Immunologic Response Rate)
Description: An Enzyme-Linked Immunosorbent Spot (ELISPOT) assay was planned to be used to demonstrate a cell mediated immune response to V935 and/or V934 in vaccinated participants. Collection of Peripheral Blood Mononuclear Cells (PBMCs) and serum took place at baseline (Screening and pre-vaccination Day 1), and various time points post vaccination across the three distinct regimens to be tested. A positive immune response was to be defined by a minimum number of spot-forming cells per million PBMC (SFC/10^6 PBMCs) for the antigen well and a minimum n-fold increase in the antigen well over the control well.
Time Frame: From pre-vaccination to Week 69
Population: Planned analysis for the secondary endpoint of Immunologic Response Rate was not performed due to study de-prioritization.
Groups:
- Part B: V935 LD/V934 Booster: Participants who completed Part A could enter Part B. Following a 12-week observation, 3 EP injections of V934 booster were administered, 1 given every 2 weeks.
- Part B: V935 HD/V934 Booster: Participants who completed Part A could enter Part B. Following a 12-week observation period, V934-EP booster was administered, 1 given every 2 weeks for 3 doses.
Arm/Group | Part A: V935 LD | Part A: V934 LD(3)+V935 LD | Part A: V935 HD | Part A: V934 HD(3)+V935 HD | Part A: V934 HD(5)+V935 HD | Part B: V935 LD/V934 Booster | Part B: V934 LD(3)+V935 LD/V934 Booster | Part B: V935 HD/V934 Booster | Part B: V934 HD(3)+V935 HD/V934 Booster | Part B: V934 HD(5)+V935 HD/V934 Booster
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs reported for Treatment Period+Acute FU+Chronic FU;Part A: Day 1 up to Wk 69, Part B: Day 1 up to 6 months post last vaccination-Wk 28). Nonserious AEs (Parts A&B) reported for Treatment Period+Acute FU;Day 1 up to 30 days post last vaccination-77 Wks
Description: Participants who completed Part A had the option to enter Part B.
Arm/Group | Part A: V935 LD | Part A: V934 LD(3)+V935 LD | Part A: V935 HD | Part A: V934 HD(3)+V935 HD | Part A: V934 HD(5)+V935 HD | Part B: V935 LD/V934 Booster | Part B: V934 LD(3)+V935 LD/V934 Booster | Part B: V935 HD/V934 Booster | Part B: V934 HD(3)+V935 HD/V934 Booster | Part B: V934 HD(5)+V935 HD/V934 Booster
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/10 | 2/11 | 1/10 | 0/1 | 0/2 | 0/7 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/10 | 11/11 | 10/10 | 1/1 | 1/2 | 3/7 | 8/9 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: V935 LD (N=3) | Part A: V934 LD(3)+V935 LD (N=3) | Part A: V935 HD (N=10) | Part A: V934 HD(3)+V935 HD (N=11) | Part A: V934 HD(5)+V935 HD (N=10) | Part B: V935 LD/V934 Booster (N=1) | Part B: V934 LD(3)+V935 LD/V934 Booster (N=2) | Part B: V935 HD/V934 Booster (N=7) | Part B: V934 HD(3)+V935 HD/V934 Booster (N=9) | Part B: V934 HD(5)+V935 HD/V934 Booster (N=9)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: V935 LD (N=3) | Part A: V934 LD(3)+V935 LD (N=3) | Part A: V935 HD (N=10) | Part A: V934 HD(3)+V935 HD (N=11) | Part A: V934 HD(5)+V935 HD (N=10) | Part B: V935 LD/V934 Booster (N=1) | Part B: V934 LD(3)+V935 LD/V934 Booster (N=2) | Part B: V935 HD/V934 Booster (N=7) | Part B: V934 HD(3)+V935 HD/V934 Booster (N=9) | Part B: V934 HD(5)+V935 HD/V934 Booster (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (11) | 6 (10) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (3) | 0 (0) | 8 (19) | 6 (17) | 0 (0) | 0 (0) | 1 (3) | 6 (11) | 3 (6)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 8 (21) | 9 (38) | 1 (1) | 1 (1) | 3 (7) | 5 (12) | 7 (14)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site scab (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site scar (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (13) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 4 (6) | 2 (2)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Celllulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear lobe infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mountain sickness acute (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.